CLINICAL TRIAL: NCT01084837
Title: A National, Multicentric, Open-label Study of Induction Treatment With VELCADE and Dexamethasone for Previously Untreated Patients With Multiple Myeloma and Renal Failure
Brief Title: Study of Induction Treatment With Velcade and Dexamethasone for Previously Untreated Patients With Multiple Myeloma and Renal Failure
Acronym: RENVEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RENVEL
Record Dates: First submitted 2010-03-07; First posted 2010-03-11 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Renal failure
MeSH Terms: conditions — Multiple Myeloma; Renal Insufficiency | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: velcade — INDUCTIoN (Cycles 1-4)
  * Bortezomib 1,3 mg/m2 i.v. days 1, 4, 8 and 11 follow by 10 days without treatment
  * Dexamethasone 40 mg/p.o. days 1-4 and 9-12 cycles 1-4 (Cycles of 21 days)
  For patients wich is not planned autotransplantation, add:
  Cycles 5-8
  * Bortezomib 1,3 mg/m2 i.v. days 1, 4, 8 and 11 follow by 10 days without treatment
  * Dexamethasone 40 mg/v.o. days 1-4 (Cycles of 21 days)
  EXTENSION TREATMENT(Cycles 9-12)
  * Bortezomib 1,3 mg/m2 i.v. days 1, 8, 15 and 22
  * Dexamethasone 40 mg/d v.o. days 1-4 (Every 6 weeks)

SUMMARY:
Primary outcome measure:

* Analyze the efficacy (in order to evaluate the response) of Bortezomib/Dexamethasone treatment

Secondary outcome measures:

* Study the speed of response and the response rate (M component in serum and urine protein) after each bortezomib/dexamethasone cycle
* Compare the efficacy of the bortezomib/dexamethasone therapy against the therapy without bortezomib
* Reversibility of renal failure
* Predictive value in the light chain determination for response and reversibility of renal failure
* Early morbidity (< 2 months)
* Progression-free survival
* Overall survival

The safety outcome consists in:

* Determining the safety and tolerance of VELCADE/Dexamethasone, according to the toxicity criteria of clinical and laboratory events

DETAILED DESCRIPTION:
60 patients, 18 years or older, diagnosed with newly symptomatic multiple myeloma (standard diagnosis criteria) and renal failure, previously untreated with chemotherapy, will be included.

It is an multi centric, national and open study designed in order to determine efficacy of the combination of bortezomib and dexamethasone for multiple myeloma patients with renal failure.

The trial consists of two parts: pre-treatment and treatment. Pre- treatment phase: include the enrolment visit in order to determine that the patient is eligible to participate in a study. The patient will be given the Informed Consent Form in order to participate in the study, and detailed information about the treatment, its benefits and risks.

Treatment phase: include the treatment which consist of, at the most, 12 cycles of Velcade and Dexamethasone (induction and extension). During these periods, patients will come to the centre for the study visits to be evaluated, the days they will receive Velcade® of each cycle.

Once the clinical trial has finished, patients will be monitored during short and long-term periods where progression free survival and overall survival will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The patient must, according with investigator criteria, be able to comply with all the protocol requirements
* The patient or legal representative must sign voluntarily the informed consent before the performance of any study related procedure, not part of usual medical care, with the knowledge that can leave the study the moment he/she wants, without prejudice to later medical care
* 18 years and older
* Patients with newly diagnosed symptomatic multiple myeloma43 which hasn't been treated previously with any chemotherapy used for this disease (see Annex 8)
* Patient with a measurable or evaluable disease, defined as follows:

  * For secretor multiple myeloma, measurable disease is defined as any quantifiable serum monoclonal protein value of IgG>10g/l or IgA > 5 g/l and, where applicable, urine light-chain excretion of ≥ 200 mg/24 hours
  * For oligo or non-secretor multiple myeloma, measurable disease is defined by the presence of soft tissue plasmocytomas (not bone) determined by clinical examination or applicable radiographs (i.e. MRI, CT-Scan). In patients with low secretor multiple myeloma, the serum and/or urine M-protein measurements are very low and difficult to follow for response assessment. In patients with non-secretor multiple myeloma, there is no M-protein in serum or urine by immunofixation
* ECOG performance status ≤ 2 (see Appendix 5)
* Patient has a life-expectancy >3 months
* Glomerular filtration calculated with MDRD <50 ml/min
* Patient has the following laboratory values during the 14 days before first dose:

  * Platelet count ≥ 50x109/l
  * Absolute neutrophil count (ANC) ≥ 0.75 x 10 9/ L
  * Corrected serum calcium (see Appendix 15) ≤ 14mg/dl
  * Aspartate transaminase (AST): ≤ 2,5 x upper limit of normal
  * Alanine Aminotransferase (ALT): ≤ 2,5 x upper limit of normal
  * Total bilirubin: ≤ 1,5 x upper limit of normal

Exclusion Criteria:

* Glomerular filtration calculated with MDRD ≥ 50ml/min
* Asymptomatic MM with renal failure from unrelated causes
* Prior Velcade therapy
* Patients previously received treatment to Multiple Myeloma
* Patient had major surgery within 4 weeks previous inclusion
* Patient with platelet count ≤ 50 x 109/l within 14 days before enrolment
* Patient with absolute neutrophil count ≤ 0,75x109/l within 14 days before enrolment
* Patients with Grade 2 peripheral neuropathy within 14 days before enrolment
* Patient has hypersensitivity to bortezomib, boron or mannitol
* Patient has received other investigational drugs within 14 days before enrolment
* Patient is known to be seropositive for the human immunodeficiency virus (HIV)
* Patient had a myocardial infarction within 6 months before of enrolment or has Class III or IV heart failure (New York Heart Association <NYHA>), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiography evidence of acute ischemia or active conduction system abnormalities, or other heart condition which, according with the specialist, can result in heart failure
* Patient is enrolled in another clinical research study and/or is receiving an investigational agent for any reason
* Patients with diffuse pulmonary disease and/or pericardial disease
* Pregnancy or breast-feed women and women of childbearing age that don't accept to use anticonceptive methods since beginning during all the study until 30 days after last cycle treatment. Fertile male patients must use effective form of contraception since enrolment, during and until 30 days after last cycle study treatment
* Patient with a previous clinical history of another malign illness except for squamous cell carcinoma or skin cancer or cervical or breast cancer) except the patient could be free of symptoms during ≥ 5 years
* Uncontrolled arterial hypertension or diabetes mellitus or other serious medical condition which places the subject at unacceptable risk or other psychiatric illness that would prevent the subject from understanding the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2012-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Efficacy | 2 years
  Analyze the efficacy (in order to evaluate the response) of Bortezomib/Dexamethasone treatment

SECONDARY OUTCOMES:
Progression-free survival | 2 years
Overall survival | 4 years
Safety | 1 year
  Determining the safety and tolerance of VELCADE/Dexamethasone, according to the toxicity criteria of clinical and laboratory events

CONTACTS AND LOCATIONS:
Locations (11):
- Spain (11):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clinic, Barcelona, Barcelona
  - Hospital de Sant Pau, Barcelona, Barcelona
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario, Salamanca, Salamanca
  - Hospital General, Segovia, Segovia
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Tenerife
  - Hospital La Fe, Valencia, Valencia
  - Hospital Lozano Blesa, Zaragoza, Zaragoza

REFERENCES:
- See also: web Haematology Spanish Association — http://aehh.org